CLINICAL TRIAL: NCT01095458
Title: Equivalent Weight Loss for Phone and Clinic Weight Management Programs
Brief Title: Phone Versus Clinical Approach to Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSCL16529; R01DK076063 (NIH)
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Obesity
Keywords: Obesity; Phone vs Clinical methods
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phone based weight management group (Experimental): Group based weight management program delivered via conference calls
  Interventions: Behavioral: Phone versus Clinic Weight Management Programs
- Clinic based weight management group (Experimental): Traditional clinical based group weight management program
  Interventions: Behavioral: Phone versus Clinic Weight Management Programs

INTERVENTIONS:
Behavioral: Phone versus Clinic Weight Management Programs — To determine if weight loss is equivalent between individuals that complete weight loss meetings in person versus on the phone.
  Other Names: Phone based weight management; Clinic based weight management

SUMMARY:
Weight loss and maintenance continues to be problematic for individuals who are overweight or obese. State-of-the-art treatment generally involves a behavioral weight loss clinic that emphasizes nutrition, physical activity, and lifestyle changes and is delivered face-to-face between health educators and small groups of participants. This delivery system is time consuming, expensive, and presents numerous barriers to the participant. We have developed a phone based delivery system that eliminates many of these barriers by substituting group conference calls for clinics and by delivering weight loss materials and products directly to the participant.

Hypothesis 1: We expect equivalent weight loss from baseline for phone and clinic groups and have defined equivalence as no greater than 4 kg difference between groups based on our pilot data and potential for clinical significance.

Hypothesis 2: During weight maintenance it is likely that participants will experience some weight re-gain. We expect both phone and clinic groups to re-gain a similar amount of weight and that weight for both groups at 18 months will be significantly less than baseline weights.

Hypothesis 3: We will complete a cost analysis to determine which delivery method is more economical. Specifically, we expect the phone delivery system to be more cost effective than that of the in-person clinics.

DETAILED DESCRIPTION:
Weight loss and maintenance continues to be problematic for individuals who are overweight or obese. State-of-the-art treatment is delivered face-to-face between care providers and small groups of participants and this is time consuming, expensive, and presents numerous barriers to the participant such as travel, conflict with work and home, need for child care, loss of anonymity, and others as well as the care provider such as office space, meeting rooms, inventory, etc. A pilot study of a phone based delivery system versus a traditional clinic has been completed with no difference in weight loss. The phone approach may eliminate many of the barriers of a traditional clinic by substituting conference calls for clinics and by delivering weight loss materials and products directly to the participant. In this fashion, the care provider and participants can reside in any location and receive the same information by conference phone call as that provided by clinic, and receive educational materials, weight management products, etc. by air or ground transportation.

This proposed investigation is a randomized, equivalency trial to test the effectiveness of a phone based weight management program compared to a traditional face-to-face clinic program for weight loss and weight maintenance. It is expected that at 6 months participants in the phone and clinic groups will show equivalent weight loss and that weight loss will be at least 10% lower than baseline. During weight maintenance some weight gain may occur. However, we expect both phone and clinic groups to gain a similar amount of weight and that weight for both groups at 18 months will be significantly less than baseline weights.

A formal cost analysis will be used to determine differences between phone and clinic approaches and extensive process analysis will be used to collect both qualitative and quantitative data to assess how well the programs were implemented as originally designed, challenges and barriers to effective implementation, initial and continual use of program specified activities, quality assurance measures, etc.

Relevance: If successful, the phone approach may eliminate many of the barriers inherent to the traditional face-to-face clinic, may be less expensive, and would potentially open weight management to any individual with access to a phone. We believe the likelihood of translation of this research to the public sector would seem reasonable and promising.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years,
* BMI between 25 and 39.9,
* Clearance from PCP.

Exclusion Criteria:

* Research project within previous 6 months,
* Exercise > 500 kcal/week,
* Pregnancy,
* Serious medical risk,
* Eating disorders,
* Use of special diets.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Equivalent weight loss for phone and clinic groups. | 6 months

SECONDARY OUTCOMES:
Equal weight management/regain. | 12 months
Cost Analysis | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Donnelly, EdD, Principal Investigator — University of Kansas
Locations (1):
- Energy Balance Lab, The University of Kansas, Lawrence, Kansas, United States

REFERENCES:
- [Result] Donnelly JE, Goetz J, Gibson C, Sullivan DK, Lee R, Smith BK, Lambourne K, Mayo MS, Hunt S, Lee JH, Honas JJ, Washburn RA. Equivalent weight loss for weight management programs delivered by phone and clinic. Obesity (Silver Spring). 2013 Oct;21(10):1951-9. doi: 10.1002/oby.20334. Epub 2013 May 25. PMID 23408579
- [Derived] Lambourne K, Washburn RA, Gibson C, Sullivan DK, Goetz J, Lee R, Smith BK, Mayo MS, Donnelly JE. Weight management by phone conference call: a comparison with a traditional face-to-face clinic. Rationale and design for a randomized equivalence trial. Contemp Clin Trials. 2012 Sep;33(5):1044-55. doi: 10.1016/j.cct.2012.05.014. Epub 2012 Jun 1. PMID 22664647